CLINICAL TRIAL: NCT06126614
Title: Prospective Randomized Evaluation of Emerging Novel Treatments for Infection Prophylaxis in Total Joint Replacement (PREVENT-iT)
Brief Title: Infection Prophylaxis in Total Joint Replacement
Acronym: PREVENT-iT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PiT-2023
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Periprosthetic Joint Infection
Keywords: Arthroplasty
MeSH Terms: interventions — chlorhexidine gluconate; Vancomycin; Povidone-Iodine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Povidone-Iodine 0.35% Lavage Solution (Experimental): The study lavage solution (povidone-iodine) is the final lavage and is to be poured in and left for 3 minutes then removed by suction.
  The study lavage solution will be a total volume of 1 litre, made with sterile isotonic saline.
  Interventions: Other: Povidone-Iodine
- Povidone-Iodine 0.35% Lavage Solution and Vancomycin (Experimental): The study lavage solution (povidone-iodine) is the final lavage and is to be poured in and left for 3 minutes then removed by suction. Two grams of vancomycin is applied to the deep joint (to arthrotomy in knee and deep to fascia in hip) following removal of the study lavage solution and immediately prior to closure.
  The study lavage solution will be a total volume of 1 litre, made with sterile isotonic saline.
  Interventions: Drug: Vancomycin Hydrochloride; Other: Povidone-Iodine
- Chlorhexidine Gluconate 0.05% Lavage Solution (Experimental): The study lavage solution (chlorhexidine-gluconate) is the final lavage and is to be poured in and left for 3 minutes then removed by suction.
  The study lavage solution will be a total volume of 1 litre, made with sterile isotonic saline.
  Interventions: Drug: Chlorhexidine Gluconate
- Chlorhexidine Gluconate 0.05% Lavage Solution and Vancomycin (Experimental): The study lavage solution (chlorhexidine gluconate) is the final lavage and is to be poured in and left for 3 minutes then removed by suction. Two grams of vancomycin is applied to the deep joint (to arthrotomy in knee and deep to fascia in hip) following removal of the study lavage solution and immediately prior to closure.
  The study lavage solution will be a total volume of 1 litre, made with sterile isotonic saline.
  Interventions: Drug: Chlorhexidine Gluconate; Drug: Vancomycin Hydrochloride
- Saline Lavage Solution (Active Comparator): The study lavage solution (saline) is the final lavage and is to be poured in and left for 3 minutes then removed by suction.
  The study lavage solution will be a total volume of 1 litre.
  Interventions: Other: Saline
- Saline Lavage Solution and Vancomycin (Experimental): The study lavage solution (saline) is the final lavage and is to be poured in and left for 3 minutes then removed by suction.
  Two grams of vancomycin is applied to the deep joint (to arthrotomy in knee and deep to fascia in hip) following removal of the study lavage solution and immediately prior to closure.
  Interventions: Drug: Vancomycin Hydrochloride; Other: Saline

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — 0.05% chlorhexidine gluconate solution for irrigation
  Arms: Chlorhexidine Gluconate 0.05% Lavage Solution; Chlorhexidine Gluconate 0.05% Lavage Solution and Vancomycin
Drug: Vancomycin Hydrochloride — 2 grams of topical vancomycin hydrochloride added to the wound
  Arms: Chlorhexidine Gluconate 0.05% Lavage Solution and Vancomycin; Povidone-Iodine 0.35% Lavage Solution and Vancomycin; Saline Lavage Solution and Vancomycin
Other: Povidone-Iodine — 0.35% povidone-iodine solution for irrigation
  Arms: Povidone-Iodine 0.35% Lavage Solution; Povidone-Iodine 0.35% Lavage Solution and Vancomycin
Other: Saline — saline for irrigation
  Arms: Saline Lavage Solution; Saline Lavage Solution and Vancomycin

SUMMARY:
Osteoarthritis (OA) is the most common cause of disability in older adults worldwide affecting 7% of the global population, or more than 500 million people globally. Total joint replacements (TJR) can help bring relief to those with osteoarthritis when other treatment options are no longer helpful. Infection is the main reason hip and knee replacements "fail". Failure leads to repeat surgeries that are often more complicated and less likely to be successful than the first surgery. Reducing the risk of infection is extremely important, antiseptic washes and antibiotics may help us do that. After joint replacement surgery, orthopaedic surgeons wash and clean the surgical wound to lower the risk of infection. The goal of this clinical trial is to determine if the use of antiseptic solutions to wash the surgical site and placing an antibiotic directly into the wound will reduce the number of infections requiring reoperation. Patients having total joint replacements will be randomized (like flipping a coin) to receive 6 possible combinations of washes and / or antibiotics. Participants will be followed for one year after TJR to compare the rate of infection in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Undergoing primary or aseptic revision TJR.
3. No contraindications to study interventions.
4. Informed consent (participant or substitute decision maker) obtained and willing to comply with the protocol.

Exclusion Criteria:

1. Received antibiotics for any reason in the two weeks prior to their TJR.
2. Chronic or acute infection at or near the TJR site.
3. Prior history of periprosthetic joint infection including any reoperation due to infection.
4. Undergoing surgery for a diagnosis of a fracture.
5. Open infected wounds on affected limb.
6. Undergoing bilateral TJR.
7. Currently enrolled in a study that does not permit co-enrollment.
8. Prior enrollment in the trial including the pilot study
9. Any condition or circumstance, which in the opinion of the Investigator, interferes with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21006 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The number of reoperations due to infection | Within 1 year of total joint replacement

SECONDARY OUTCOMES:
The number of non-operative surgical site infections requiring antibiotics for treatment. | Within 1 year of total joint replacement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wood, MD, FRCSC, Principal Investigator — Hamilton Health Sciences / McMaster University
Locations (1):
- Hamilton Health Sciences - Juravinski Hospital and Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No